CLINICAL TRIAL: NCT04261075
Title: A Phase 1, First-in-Human, Multicenter, Open-label, Dose-escalation Study of IPH5201 as Monotherapy or in Combination With Durvalumab ± Oleclumab in Advanced Solid Tumors
Brief Title: IPH5201 as Monotherapy or in Combination With Durvalumab +/- Oleclumab in Subjects With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6770C00001
Record Dates: First submitted 2020-01-07; First posted 2020-02-07 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IPH5201 monotherapy dose escalation (Experimental): IPH5201 monotherapy
  Interventions: Biological: IPH5201
- IPH5201 dose escalation with durvalumab (Experimental): IPH5201 plus durvalumab
  Interventions: Biological: IPH5201; Biological: durvalumab
- IPH5201 dose escalation with durvalumab + oleclumab (Experimental): IPH5201 plus durvalumab and oleclumab
  Interventions: Biological: IPH5201; Biological: durvalumab; Biological: oleclumab

INTERVENTIONS:
Biological: IPH5201 — Ascending dose levels of IPH5201 every 3 weeks (Q3W) for a maximum of 2 years
Biological: durvalumab — Durvalumab Q3W for a maximum of 2 years
  Arms: IPH5201 dose escalation with durvalumab; IPH5201 dose escalation with durvalumab + oleclumab
Biological: oleclumab — Oleclumab Q3W for a maximum of 2 years
  Arms: IPH5201 dose escalation with durvalumab + oleclumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability and to determine the dose of IPH5201 that can be used as monotherapy or in combination with durvalumab +/- oleclumab in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Study D6770C00001 is a Phase 1, first-in-human, multicenter, open-label, dose-escalation study to evaluate the safety, tolerability, antitumor activity, pharmacokinetics, and immunogenicity of IPH5201 in adult subjects with advanced solid tumors, when administered as monotherapy or in combination with durvalumab ± oleclumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects; age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Subjects diagnosed with advanced solid tumors.
* For Part 1 and Part 2 (IPH5201 in monotherapy or combined with durvalumab):Subjects must be refractory to standard therapy or for which no standard therapy exists.
* For Part 3 (IPH5201 combined with durvalumab and oleclumab): Subjects must have received and radiologically progressed on 1 prior line of systemic therapy for metastatic pancreatic ductal adenocarcinoma.
* Subjects must have at least 1 measurable lesion according to RECIST v1.1.
* Subjects must provide tumor specimens .

Exclusion Criteria:

* Receipt of any conventional or investigational anticancer therapy (anti-CTLA-4, anti-PD-1, anti-PD-L1 antibodies) within 21 days of the planned first dose.
* Receipt of agents targeting CD73, CD39, or adenosine receptors.
* Concurrent enrollment in another therapeutic clinical study.
* Any toxicity (excluding alopecia) from prior standard therapy that has not been completely resolved to baseline at the time of consent.

  * No toxicity leading to permanent discontinuation of prior IO therapy
  * Subjects must not have required the use of additional immunosuppression other than corticosteroids
* Active or prior documented autoimmune or inflammatory disorders within the past 5 years
* Cardiac and vascular criteria:

  * Presence of myocardial infarction or unstable angina , or stroke, within 6 months.
  * Congestive heart failure, serious cardiac arrhythmia requiring medication, or uncontrolled hypertension
  * History of severe hypertension
  * History of any grade of blood clot within 6 months
* Active infection, including tuberculosis; hepatitis B virus (HBV); hepatitis C virus (HCV); or human immunodeficiency virus (HIV)
* Uncontrolled illness including certain lung diseases, uncontrolled diabetes, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study.
* Other invasive malignancy within 2 years.
* Major surgery within 28 days prior to first dose
* Female subjects who are pregnant or breast feeding

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as a measure of safety | From time of informed consent through treatment period and including the follow-up 12 weeks after last dose of investigational product, approximately 7 months
  The primary endpoint is safety as assessed by the presence of adverse events (AEs), serious adverse events (SAEs), and dose limiting toxicities (DLTs).
Incidence of clinically significant laboratory values as a measure of safety | From time of informed consent through 12 weeks after the last dose of investigational product, approximately 7 months
  Number of subjects with clinically significant laboratory values from baseline including blood counts, liver, kidney and pancreas tests, electrolytes, and blood clotting.
Incidence of clinically significant electrocardiogram (ECG) abnormalities as a measure of safety | From time of informed consent through treatment period and including the follow-up period 12 weeks after last dose of investigational product, approximatley 7 months
  12 lead ECGs will be measured to identify clinical significant abnormalities including ECGs that demonstrate a QTcF value >500ms, 2 additional 12-lead ECGs should be obtained over a 30 minute time period to confirm prolongation based on the average QTcF value

SECONDARY OUTCOMES:
OR (Objective Response; Response evaluation criteria in solid tumors [RECIST] v1.1) | From time of consent until date of first documented disease progression (approximately 4 months)
  Evaluate the primary antitumor activity of IPH5201 monotherapy or in combination with durvalumab +/- oleclumab (disease control)
DC (Disease Control; RECIST 1.1) | From time of consent until date of first documented disease progression (approximately 4 months)
  Evaluate the primary antitumor activity of IPH5201 with durvalumab +/- oleclumab (disease control)
Half-life of IPH5201 | From start of treatment through Cycle 6 (21 day cycle, approximately 5 months)
  To characterize the pharmacokinetics of IPH5201 as monotherapy and in combination with durvalumab ± oleclumab
Maximum serum concentration (Cmax) of IPH5201 | From start of treatment through Cycle 6 (21 day cycle, approximately 5 months)
  To characterize the pharmacokinetics of IPH5201 as monotherapy and in combination with durvalumab ± oleclumab
Area under the curve (AUC) of IPH5201 | From start of treatment through Cycle 6 (21 day cycle, approximately 5 months)
  To characterize the pharmacokinetics of IPH5201 as monotherapy and in combination with durvalumab ± oleclumab
Serum trough concentrations (durvalumab) | From start of treatment through Cycle 6 (21 day cycle, approximately 5 months)
  To determine the pharmacokinetics of durvalumab when administered in combination with IPH5201+/- oleclumab
Serum trough concentrations (oleclumab) | From start of treatment through Cycle 6 (21 day cycle, approximately 5 months)
  To determine the pharmacokinetics of oleclumab in combination with durvalumab and IPH5201
Incidence of antidrug antibodies (IPH5201) | From start of treatment until 90 days after end of treatment (approximately 7 months)
  To determine the immunogenicity of IPH5201 as monotherapy and in combination with durvalumab ± oleclumab
Incidence of antidrug antibodies (durvalumab) | From start of treatment until 90 days after end of treatment (approximately 7 months)
  To determine the immunogenicity of durvalumab in combination with IPH5201 ± oleclumab
Incidence of antidrug antibodies (oleclumab) | From start of treatment until 90 days after end of treatment (approximately 7 months)
  To determine the immunogenicity of oleclumab in combination with IPH5201 + durvalumab

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Research Site, Huntersville, North Carolina
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
- France (2):
  - Research Site, Bordeaux
  - Research Site, Villejuif
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No